CLINICAL TRIAL: NCT06596525
Title: Effects of Barefoot vs. Shod Whole Body Vibration Training on Pedobarographic Evaluation, Balance, Endurance and Lower Extremity Functions in Children With Cerebral Palsy: 3-Arm Randomized Controlled Single-Blind Study
Brief Title: Effects of Barefoot vs. Shod Whole Body Vibration Training in Children With Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, FİLİZ TUNA, Assoc. Prof., Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUTF-GOBAEK 2024/322
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy; whole body vibration; conventional physical therapy; balance; pedobarographic evaluation; gross motor function; spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a single-blind randomized controlled trial with 3 parallel arms, including 2 experimental groups and 1 control group. Participants will be randomized into 3 groups at the beginning of the study.
  One arm (Group 1) will be sham comparator and will receive sham WBVT in addition to conventional physical therapy. The other two arms are the experimental groups. Group 2 will receive WBVT with footwear in addition to conventional physical therapy, and Group 3 will receive WBVT with barefoot in addition to conventional physical therapy.
  Group 1:Conventional physical therapy (PT) + WBVTsh (sham)
  Group 2: PT + WBVTs (shod)
  Group 3: PT+ WBVTb (barefoot)
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to study groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Conventional physical therapy (PT) + WBVTsh (sham) (Sham Comparator): Group 1 will receive a "sham" WBVT in addition to conventional physical therapy. Over a period of 4 weeks, 3 days per week for 30 minutes each session, participants will engage in conventional physical therapy program.
  Interventions: Other: Conventional physical therapy; Other: Sham Whole Body Vibration Training (WBVTsh)
- Group 2: Conventional physical therapy (PT) + WBVTs (shod) (Experimental): Over a period of 4 weeks, in addition to conventional physical therapy program, the participants will engage in WBVT on commercially available "ThinningPlate" vibration platform, 3 days per week for 15 minutes each session. Group 2 will wear everyday sports shoes during WBVT.
  Interventions: Other: Conventional physical therapy; Other: Shod Whole Body Vibration Training (WBVTs)
- Group 3: Conventional physical therapy (PT) + WBVTb (barefoot) (Experimental): Over a period of 4 weeks, in addition to conventional physical therapy program, the participants will engage in WBVT on commercially available "ThinningPlate" vibration platform, 3 days per week for 15 minutes each session. Group 3 will be barefoot during WBVT.
  Interventions: Other: Conventional physical therapy; Other: Barefoot Whole Body Vibration Training (WBVTb)

INTERVENTIONS:
Other: Conventional physical therapy — Conventional physical therapy program will include:
  1. Stretching exercises (forearm pronators, ulnar deviators, shoulder internal rotators, hip flexors and adductors, and hamstring muscle groups)
  2. Strengthening exercises (ankle dorsiflexors, knee extensors, and hip flexor muscle groups)
  3. Posture exercises
  4. Balance and proprioception exercises
  5. Walking training, obstacle crossing training, stair climbing and descending exercises
Other: Barefoot Whole Body Vibration Training (WBVTb) — Each WBVT session will consist of the following schedule: 3 minutes of WBVT- 2 minutes rest- 3 minutes of WBVT- 2 minutes rest- 3 minutes of WBVT- 2 minutes rest. Thus a treatment session will last 15 minutes in total. The participants will be barefoot. A specially designed walker will be used to provide support during WBVT for children who are unable to stand independently on the platform and. All exercises and WBVT sessions will be performed under the supervision of a physiotherapist and postural correction will be encouraged through visual feedback (the platform will be placed in front of a mirror) and verbal cueing. One set of WBVT along with the dynamic exercise program to be implemented on the platform is summarized below.
  Stage 1: Semi-squat (knees flexed 10-45º) for 1 minute
  Stage 2: Semi-squat +Calf raise for 1 minute
  Stage 3: Triceps surae stretch for 1 minute
  Arms: Group 3: Conventional physical therapy (PT) + WBVTb (barefoot)
Other: Shod Whole Body Vibration Training (WBVTs) — Each WBVT session will consist of the following schedule: 3 minutes of WBVT- 2 minutes rest- 3 minutes of WBVT- 2 minutes rest- 3 minutes of WBVT- 2 minutes rest. Thus a treatment session will last 15 minutes in total. The participants will wear everyday sports shoes. A specially designed walker will be used to provide support during WBVT for children who are unable to stand independently on the platform and. All exercises and WBVT sessions will be performed under the supervision of a physiotherapist and postural correction will be encouraged through visual feedback (the platform will be placed in front of a mirror) and verbal cueing. One set of WBVT along with the dynamic exercise program to be implemented on the platform is summarized below.
  Stage 1: Semi-squat (knees flexed 10-45º) for 1 minute
  Stage 2: Semi-squat +Calf raise for 1 minute
  Stage 3: Triceps surae stretch for 1 minute
  Arms: Group 2: Conventional physical therapy (PT) + WBVTs (shod)
Other: Sham Whole Body Vibration Training (WBVTsh) — During "Sham" WBVT; the same exercises that the intervention groups will receive on the vibration platform will be performed on the platform for the same duration (3 days per week for 15 minutes each session, over a period of 4 weeks) without the platform being activated.
  Arms: Group 1: Conventional physical therapy (PT) + WBVTsh (sham)

SUMMARY:
Cerebral palsy (CP) refers to a group of lifelong conditions that affect the development of movement and coordination that lead to activity limitations due to damage to the developing fetal or neonatal brain tissue. Although the brain lesion is static, it can lead to progressive musculoskeletal system problems. As a result of the restriction of ankle joint range of motion and many microscopic changes in the muscle structure, plantar pressure distribution is impaired in children with CP which brings about gait and balance problems. Moreover, since physical activity may be restricted due to spasticity, poor motor control, muscle weakness and balance problems; the main goals in CP rehabilitation are normalization of muscle tone, improving walking function by increasing joint range of motion, strength and balance and consequently improving mobility.

There is a need for adjunctive treatment methods with low side effect profiles that can be applied in the long term to prevent musculoskeletal complications and preserve existing functions in children with CP. Whole body vibration training (WBVT), is a therapeutic exercise method that is growing in popularity due to its ease of application, low side effect profile and non-invasiveness as an auxiliary treatment method to traditional rehabilitation programs. Although WBVT is suggested as an easily applicable and safe treatment method with home-type vibration devices; scientific evidence is still lacking and it has not yet been included in routine rehabilitation programs due to the small number of high-quality randomized controlled trials. This study aims to determine the efficacy of barefoot vs. shod WBVT in addition to the conventional physiotherapy, compared to the conventional physiotherapy alone, in children with mild-moderate CP on pedobarographic evaluation, balance, endurance and lower extremity functions. As a result of this study, it might possible to offer children with CP an accessible, safe and helpful treatment method with established protocols.

DETAILED DESCRIPTION:
CP describes a group of neurological disorders that occur after damage to the brain during development. Although brain damage is non-progressive; spasticity, poor motor control, muscle weakness and balance problems are frequently observed due to first motor neuron damage. Restriction of physical activity causes joint contractures and bone deformities, which negatively affect muscle strength and motor function. The main goals in CP treatment are to normalize muscle tone, reduce joint stiffness, increase joint range of motion, strength and balance.

In children with CP, while proximal motor function of the lower extremities is generally preserved; calf muscles, which are well-known to greatly influence postural control, are particularly affected by primary impairments such as spasticity, selective motor control deficits and weakness. As gastrocnemius muscle stiffness increases with growth, it undergoes shortening and atrophy; while its antagonist muscle, the tibialis anterior, often becomes weak. In later ages, ankle joint of motion progressively decreases, accompanied by numerous microscopic changes in muscle structure leading to plantar flexion contractures in children with CP. This results in abnormal plantar pressure distribution, contributing to gait and balance problems. Increased plantar flexor activity or knee flexion increases load on the forefoot. Significant differences have been reported in weight distribution on the feet of children with hemiplegic CP. Previous studies suggest that children with CP exhibit distinct plantar pressure patterns.

WBVT is an emerging therapeutic exercise method in addition to traditional rehabilitation, gaining popularity due to its ease of application and low side effect profile. In WBVT, vibration motion generated by the platform stimulates a movement pattern similar to human gait which results in activation of proprioceptive spinal circuits, leading to compensatory rhythmic muscle contractions in the lower extremities and trunk. Studies conducted on adult, adolescent and pediatric individuals with CP report positive effects of WBVT on gross motor function, balance, muscle strength, muscle tone, spasticity, proprioceptive perception, functional activities and walking. In brief, WBVT stands out as a safe, non-pharmacological method to increase muscle mass in specific pediatric populations.

Enhancing balance and lower extremity function is crucial for improving mobilization, a key goal in CP treatment. CP is commonly approached as a pediatric issue, but approximately 90% of individuals with CP reach adulthood and their life expectancy is similar to that of general population. Given that CP is a lifelong condition, there is a need for adjunctive therapies with low side effect profiles that can be applied in the long term to prevent complications and preserve existing functions. WBVT emerges as a promising adjunctive therapy for inclusion in rehabilitation programs for CP. It is non-invasive, easy to administer and has low side effect profile. WBVT can be applied quickly and conveniently with home-based devices, making it a practical treatment option.

Not only is the number of randomized controlled trials limited, but existing studies also have shortcomings such as a lack of specification regarding footwear (shoes/socks/barefoot/assistive devices) used during WBVT, as well as addressing technical terms (frequency, peak-to-peak displacement, amplitude, etc.), type of vibration (side alternating/synchronous), and the types of exercises (static or dynamic) performed on the platform.

In this study, participants will be selected from children diagnosed with CP who are followed up at the pediatric rehabilitation clinic of Trakya University Department of Physical Medicine and Rehabilitation and who meet the inclusion and exclusion criteria. Participants will be randomized into 3 groups at the beginning of the study. Age, gender, more affected extremity, use of orthoses/assistive devices, Gross Motor Function Classification System (GMFCS) level, history of orthopedic surgery and presence of comorbidities will be recorded for all participants. Written informed consent will be obtained from the families of all participants.

Group 1 will receive sham WBVT in addition to conventional physical therapy program. Groups 2 and 3 will receive WBVT with footwear and barefoot, respectively in addition to conventional physical therapy program. This study aims to determine the efficacy of barefoot vs. shod WBVT in addition to the conventional physiotherapy, compared to the conventional physiotherapy alone, in children with mild-moderate CP on pedobarographic evaluation, balance, endurance and lower extremity functions. By addressing the gaps in the literature and establishing the effects of WBVT, it is anticipated that WBVT will contribute to improving mobility, balance and overall quality of life for children with CP. Detailed protocol presentation in this study will contribute to pediatric rehabilitation in clinical practice and shed light on future research.

ELIGIBILITY:
Inclusion Criteria:

1. Between ages of 3 and 18
2. Diagnosed with CP
3. Able to walk at least 10 meters with or without assistive devices
4. GMFCS level 1-3
5. Able to stand independently or with self-support on a vibration platform for 3 minutes
6. Able to understand verbal commands and cooperate during clinical examination

Exclusion Criteria:

1. History of lower extremity botulinum toxin injection or surgery in the past 6 months
2. Any bone fracture in the past 8 weeks
3. Acute thrombosis, muscle-tendon inflammation, nephrolithiasis
4. Presence of implants in the spine or lower extremities
5. Pregnancy
6. Presence of mental impairment, visual or hearing loss affecting balance
7. History of seizures in the past 6 months
8. ASH 4 spasticity/contracture in any lower extremity muscle group
9. Presence of cardiovascular or pulmonary disease
10. Diagnosis of dyskinetic cerebral palsy

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pedobarographic evaluation | At baseline, at the end of the 4-week treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  Static and dynamic plantar pressure parameters will be recorded via pedobarographic evaluation platform. All analysis will be carried out on a flat platform at a constant temperature of 18-22 degrees. All participants will receive clear instructions on test protocols and will be recommended to dress in a way that does not impede lower extremity movements.
Balance | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week).
  Bipedal, unipedal and sitting balance will be evaluated using balance plates.

SECONDARY OUTCOMES:
Bioimpedance analysis | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  TANİTA MC 780 multi-frequency segmental body composition analyzer will be used for the assessment.
Modified Ashworth Scale (MAS) for lower extremity muscle tone | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  For clinical assessment of spasticity of lower extremity muscles, the Modified Ashworth Scale (MAS) will be used. It is based on the subjective grading of resistance felt during examination. MAS grades range from 0 (normal muscle tone) to 4 (extreme spasticity).
Pediatric Balance Scale (PBS) | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  The Pediatric Balance Scale (PBS) is a highly reliable scale in children with CP and will be used to assess functional balance of the participants. The PBS is an adaptation for children by Franjoine of the Berg Balance Scale. It includes functional movements such as sitting, standing up, transferring, standing on one foot, and picking up objects from the ground, comprising 14 sections scored from 0 to 4 each; the maximum score achievable is 56.
Timed up and go (TUG) test | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  Functional mobility of the participants will be evaluated through timed up and go (TUG) test. TUG test is a test that evaluates the balance function of an individual during basic mobility. The patient is asked to rise from a chair without using their arms for support, walk at their maximum safe speed for a distance of 3 meters (approximately 10 feet), turn around, return to the chair, and sit down again. This process is repeated three times, and the time taken to complete the task is recorded in seconds. A shorter time indicates better balance performance.
Lower extremity muscle strength | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  Lower extremity muscle strength will ve evaluated through Medical Research Council (MRC) Scale, which provides a standardized method to quantify muscle strength based on observed movement against resistance. The MRC Scale categorizes muscle strength into grades from 0 to 5: 0 (no contraction), 1 (trace contraction, muscle flicker, but no movement), 2 (active movement with gravity eliminated), 3 (active movement against gravity), 4 (active movement against some resistance), 5 (normal strength, movement against full resistance).
Five times sit-to-stand test (5XSST) | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  Five times sit-to-stand test (5XSST) will be used to assess lower extremity functional strength and balance. The participant begins the test sitting on the chair with arms crossed over the chest. They are instructed to stand up and sit down from the chair five times as quickly as possible without using arm support. The lowest time recorded from two trials is used as the final score.
Gross Motor Function Measure (GMFM-88) | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  Gross Motor Function Measure (GMFM-88) is a standardized observational test designed to measure changes in gross motor function in children with CP. It has 5 dimensions of interest: A: Lying and rolling, B: Sitting, C: Crawling and kneeling, D: Standing, E: Walking, running and jumping. A scoring key of 0 (does not initiate), 1 (initiates), 2 (partially completes), 3 (completed) is used; however the parameters such as distance, time, support provided, accuracy, counts and tasks will determine the specific item scores. Item scores are summed to calculate raw and percent scores fro each of the five GMFM-88 dimensions. Dimension percent scores are averaged to obtain an overall total score. Not tested items in the GMFM-88 are scored as "0".
6 minutes walk test | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  6-minute walk test will be used to assess the participant's functional status and endurance. It provides an indirect assessment of an individual's capacity during daily life activities and can also be used to monitor progress during treatment. It measures the distance a patient can walk on a flat, hard surface at their maximum speed over a period of 6 minutes. This time-based test is conducted in quiet and enclosed corridors, recording parameters such as effort expended over a specific time period, oxygen saturation, heart rate, blood pressure, respiratory rate, and walking distance.
Functional mobility scale (FMS) | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  The FMS classifies the functional mobility of children 4-18 years of age with cerebral palsy, taking into account the assistive devices a child might use. Higher scores mean better outcome.
The Gillette Functional Assessment Questionnaire (FAQ) | At baseline, after the end of the treatment (at 4th week), 1 month after the end of treatment (at 8th week)
  The Gillette Functional Assessment Questionnaire (FAQ) is a self or proxy-report measure that includes a ten-level classification of ambulatory function (FAQ Walking Scale), and 22 functional locomotor activities rated on a five-level Likert difficulty scale (FAQ 22-item skill set). The FAQ is intended for use in individuals with all levels of walking ability, and focuses on what an individual can do independently with the use of assistive devices or orthoses as needed to maximize function.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Tuna, Assoc. Prof, Principal Investigator — Trakya University; Nur Kakilli, M.D., Principal Investigator — Trakya University
Locations (1):
- Trakya University Faculty of Medicine, Edirne, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruck J, Chabot G, Rauch F. Vibration treatment in cerebral palsy: A randomized controlled pilot study. J Musculoskelet Neuronal Interact. 2010 Mar;10(1):77-83. PMID 20190383
- [Background] Leite HR, Camargos ACR, Mendonca VA, Lacerda ACR, Soares BA, Oliveira VC. Current evidence does not support whole body vibration in clinical practice in children and adolescents with disabilities: a systematic review of randomized controlled trial. Braz J Phys Ther. 2019 May-Jun;23(3):196-211. doi: 10.1016/j.bjpt.2018.09.005. Epub 2018 Sep 19. PMID 30245042
- [Background] Sa-Caputo DC, Costa-Cavalcanti R, Carvalho-Lima RP, Arnobio A, Bernardo RM, Ronikeile-Costa P, Kutter C, Giehl PM, Asad NR, Paiva DN, Pereira HV, Unger M, Marin PJ, Bernardo-Filho M. Systematic review of whole body vibration exercises in the treatment of cerebral palsy: Brief report. Dev Neurorehabil. 2016 Oct;19(5):327-33. doi: 10.3109/17518423.2014.994713. Epub 2015 Mar 31. PMID 25826535
- [Background] Young NL. The transition to adulthood for children with cerebral palsy: what do we know about their health care needs? J Pediatr Orthop. 2007 Jun;27(4):476-9. doi: 10.1097/01.bpb.0000271311.87997.e7. No abstract available. PMID 17513974
- [Background] Rauch F, Sievanen H, Boonen S, Cardinale M, Degens H, Felsenberg D, Roth J, Schoenau E, Verschueren S, Rittweger J; International Society of Musculoskeletal and Neuronal Interactions. Reporting whole-body vibration intervention studies: recommendations of the International Society of Musculoskeletal and Neuronal Interactions. J Musculoskelet Neuronal Interact. 2010 Sep;10(3):193-8. PMID 20811143
- [Background] Swolin-Eide D, Magnusson P. Does Whole-Body Vibration Treatment Make Children's Bones Stronger? Curr Osteoporos Rep. 2020 Oct;18(5):471-479. doi: 10.1007/s11914-020-00608-0. PMID 32696294
- [Background] Tekin F, Kavlak E. Short and Long-Term Effects of Whole-Body Vibration on Spasticity and Motor Performance in Children With Hemiparetic Cerebral Palsy. Percept Mot Skills. 2021 Jun;128(3):1107-1129. doi: 10.1177/0031512521991095. Epub 2021 Feb 3. PMID 33535899
- [Background] Martakis K, Stark C, Rehberg M, Semler O, Duran I, Schoenau E. Reference Centiles to Monitor the 6-minute-walk Test in Ambulant Children with Cerebral Palsy and Identification of Effects after Rehabilitation Utilizing Whole-body Vibration. Dev Neurorehabil. 2021 Jan;24(1):45-55. doi: 10.1080/17518423.2020.1770891. Epub 2020 Jun 21. PMID 32564635
- [Background] Wren TA, Lee DC, Hara R, Rethlefsen SA, Kay RM, Dorey FJ, Gilsanz V. Effect of high-frequency, low-magnitude vibration on bone and muscle in children with cerebral palsy. J Pediatr Orthop. 2010 Oct-Nov;30(7):732-8. doi: 10.1097/BPO.0b013e3181efbabc. PMID 20864862
- [Background] Ko MS, Sim YJ, Kim DH, Jeon HS. Effects of Three Weeks of Whole-Body Vibration Training on Joint-Position Sense, Balance, and Gait in Children with Cerebral Palsy: A Randomized Controlled Study. Physiother Can. 2016;68(2):99-105. doi: 10.3138/ptc.2014-77. PMID 27909356
- [Background] Tupimai T, Peungsuwan P, Prasertnoo J, Yamauchi J. Effect of combining passive muscle stretching and whole body vibration on spasticity and physical performance of children and adolescents with cerebral palsy. J Phys Ther Sci. 2016 Jan;28(1):7-13. doi: 10.1589/jpts.28.7. Epub 2016 Jan 30. PMID 26957720
- [Background] El-Shamy SM. Effect of whole-body vibration on muscle strength and balance in diplegic cerebral palsy: a randomized controlled trial. Am J Phys Med Rehabil. 2014 Feb;93(2):114-21. doi: 10.1097/PHM.0b013e3182a541a4. PMID 24434887
- [Background] Ahlborg L, Andersson C, Julin P. Whole-body vibration training compared with resistance training: effect on spasticity, muscle strength and motor performance in adults with cerebral palsy. J Rehabil Med. 2006 Sep;38(5):302-8. doi: 10.1080/16501970600680262. PMID 16931460
- [Background] Unger M, Jelsma J, Stark C. Effect of a trunk-targeted intervention using vibration on posture and gait in children with spastic type cerebral palsy: a randomized control trial. Dev Neurorehabil. 2013;16(2):79-88. doi: 10.3109/17518423.2012.715313. PMID 23477461
- [Background] Saquetto M, Carvalho V, Silva C, Conceicao C, Gomes-Neto M. The effects of whole body vibration on mobility and balance in children with cerebral palsy: a systematic review with meta-analysis. J Musculoskelet Neuronal Interact. 2015 Jun;15(2):137-44. PMID 26032205
- [Background] Matute-Llorente A, Gonzalez-Aguero A, Gomez-Cabello A, Vicente-Rodriguez G, Casajus Mallen JA. Effect of whole-body vibration therapy on health-related physical fitness in children and adolescents with disabilities: a systematic review. J Adolesc Health. 2014 Apr;54(4):385-96. doi: 10.1016/j.jadohealth.2013.11.001. Epub 2014 Jan 1. PMID 24388109
- [Background] Lopez S, Bini F, Del Percio C, Marinozzi F, Celletti C, Suppa A, Ferri R, Staltari E, Camerota F, Babiloni C. Electroencephalographic sensorimotor rhythms are modulated in the acute phase following focal vibration in healthy subjects. Neuroscience. 2017 Jun 3;352:236-248. doi: 10.1016/j.neuroscience.2017.03.015. Epub 2017 Mar 18. PMID 28323013
- [Background] Cheng HY, Yu YC, Wong AM, Tsai YS, Ju YY. Effects of an eight-week whole body vibration on lower extremity muscle tone and function in children with cerebral palsy. Res Dev Disabil. 2015 Mar;38:256-61. doi: 10.1016/j.ridd.2014.12.017. Epub 2015 Jan 7. PMID 25575288
- [Background] Schirinzi T, Romano A, Favetta M, Sancesario A, Burattini R, Summa S, Della Bella G, Castelli E, Bertini E, Petrarca M, Vasco G. Non-invasive Focal Mechanical Vibrations Delivered by Wearable Devices: An Open-Label Pilot Study in Childhood Ataxia. Front Neurol. 2018 Oct 9;9:849. doi: 10.3389/fneur.2018.00849. eCollection 2018. PMID 30356679
- [Background] Murillo N, Valls-Sole J, Vidal J, Opisso E, Medina J, Kumru H. Focal vibration in neurorehabilitation. Eur J Phys Rehabil Med. 2014 Apr;50(2):231-42. PMID 24842220
- [Background] Cochrane DJ. Vibration exercise: the potential benefits. Int J Sports Med. 2011 Feb;32(2):75-99. doi: 10.1055/s-0030-1268010. Epub 2010 Dec 16. PMID 21165804
- [Background] Galli M, Cimolin V, Pau M, Leban B, Brunner R, Albertini G. Foot pressure distribution in children with cerebral palsy while standing. Res Dev Disabil. 2015 Jun-Jul;41-42:52-7. doi: 10.1016/j.ridd.2015.05.006. Epub 2015 Jun 6. PMID 26057837
- [Background] Nsenga Leunkeu A, Lelard T, Shephard RJ, Doutrellot PL, Ahmaidi S. Gait cycle and plantar pressure distribution in children with cerebral palsy: clinically useful outcome measures for a management and rehabilitation. NeuroRehabilitation. 2014;35(4):657-63. doi: 10.3233/NRE-141163. PMID 25318772
- [Background] Femery V, Moretto P, Renaut H, Thevenon A, Lensel G. Measurement of plantar pressure distribution in hemiplegic children: changes to adaptative gait patterns in accordance with deficiency. Clin Biomech (Bristol). 2002 Jun;17(5):406-13. doi: 10.1016/s0021-9290(02)00063-5. PMID 12084546
- [Background] Wiley ME, Damiano DL. Lower-extremity strength profiles in spastic cerebral palsy. Dev Med Child Neurol. 1998 Feb;40(2):100-7. doi: 10.1111/j.1469-8749.1998.tb15369.x. PMID 9489498